CLINICAL TRIAL: NCT01185210
Title: Investigation of Alanine in Fructose Intolerance: A Randomized, Double Blind, Dose Ranging, Placebo Controlled Study
Brief Title: Investigation of Alanine in Fructose Intolerance: A Dose Ranging Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Collaborators: University of Iowa (Other); Teikyo University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fructose: Double Blind
Record Dates: First submitted 2009-09-22; First posted 2010-08-19 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Fructose Intolerance
MeSH Terms: conditions — Fructose Intolerance | interventions — Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive placebo (mix of sugar and salt).
  Interventions: Dietary Supplement: Placebo
- Alanine - 12.5 (Experimental): Subjects will receive 12.5 grams of alanine
  Interventions: Dietary Supplement: Alanine
- Alanine - 25 (Experimental): Subjects will receive 25 grams of alanine.
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects will receive placebo (mix of sugar and salt) 20 minutes before consuming fructose.
  Arms: Placebo
Dietary Supplement: Alanine — Subjects will receive 12.5 grams of alanine 20 minutes before consuming fructose.
  Arms: Alanine - 12.5
Dietary Supplement: Alanine — Subjects will receive 25 grams of alanine 20 minutes before consuming fructose.
  Arms: Alanine - 25

SUMMARY:
Background:

Over the past few decades, fructose is increasingly being used as a sweetener/ additive in a variety of foods. Incomplete absorption of fructose has been implicated as a cause of gastrointestinal symptoms. In tertiary care centers, the prevalence of fructose malabsorption in subjects with unexplained GI symptoms is thought to be between 11-50%, when assessed with breath tests following administration of 25 grams of fructose in a 10% solution. Restriction of dietary fructose has been shown to improve symptoms in these patients to an extent. Currently, there are no therapeutic agents that improve intestinal fructose absorption and thereby decrease symptoms. Studies in the pediatric population have shown that fructose absorption in the small intestine is increased in the presence of glucose or amino acids, especially alanine.

Objective:

The investigators' objective is to assess whether co-administration of an oral solution of L-alanine facilitates fructose absorption and decreases gastrointestinal (GI) symptoms associated with fructose malabsorption in subjects undergoing standard fructose breath test when compared to placebo.

Methods and analysis:

The investigators propose a randomized, double-blind study in 40 subjects with known fructose intolerance. After an overnight fast, each subject will receive an oral solution of 12.5 grams of alanine in 125cc of water or placebo. Next, the subject will receive an oral solution of 25 grams of fructose in a 10% solution. Serum, urine and breath samples will be collected at baseline and at 30-minute intervals for 4 hours. GI symptoms will also be assessed and recorded at 30 minute intervals using a standard questionnaire. Repeated measures ANOVA will be used to compare the data obtained during the study protocol with the baseline (pre-study) data.

Expected outcomes:

Co-administration of alanine with fructose may improve fructose absorption and decrease symptoms in subjects with fructose intolerance.

Hypothesis: Ingestion of alanine along with fructose, will facilitate intestinal absorption of fructose in subjects with fructose malabsorption.

Aim: To investigate the effects of co-administration of equi-molar doses of alanine on a) the absorption of fructose and b) the occurrence of GI symptoms in subjects with fructose malabsorption.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years
2. Diagnosis of fructose malabsorption (positive breath test after ingestion of 25 grams of fructose defined as either (a) ≥ 20 ppm rise of breath H2/CH4/both over baseline values or a successive rise of ≥ 5 ppm over baseline and in 3 consecutive breath samples)

Exclusion Criteria:

1. Cognitive impairment or any other inability to provide informed consent
2. Prisoners
3. GI surgery except appendectomy, cholecystectomy, caesarean section, hysterectomy
4. Antibiotics in the previous 3 months
5. Bacterial overgrowth or lactose intolerance
6. Major co-morbid illnesses, including chronic pancreatitis, celiac disease, inflammatory bowel disease, diabetes, scleroderma, pseudo-obstruction syndromes etc.
7. Known food allergies
8. Medication use: opioids, Tegaserod, laxatives, enemas
9. Diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Decrease breath Hydrogen and/or Methane production | less than 6 months

SECONDARY OUTCOMES:
Occurrence or severity of GI symptoms during the test | less than 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, Md, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States